CLINICAL TRIAL: NCT07044791
Title: Metabolic Parameters and Quality of Life in Women on Neo-/Adjuvant Therapy for Breast Cancer: a Randomized Controlled Trial on the Effectiveness of an Intensive Dietary Intervention
Brief Title: Metabolic Parameters and Quality of Life in Women on Neo-/Adjuvant Therapy for Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Grazia Arpino, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 280/17
Record Dates: First submitted 2025-05-30; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Cancer Invasive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional non-pharmacological study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: intensive nutritional intervention (Experimental): ARM A: Visits will be set up monthly in order to assess body weight, waist circumference, diet compliance (etc...) for all period of the BC adjuvant treatment (6 months).
  Interventions: Behavioral: Nutritional counseling. No drug treatment will be administered in this study.
- ARM B: standard nutritional intervention (No Intervention): ARM B: Visits will be set up only at the baseline, after 6 months namely at the end

INTERVENTIONS:
Behavioral: Nutritional counseling. No drug treatment will be administered in this study. — Nutritional counseling. No drug treatment will be administered in this study.
  Arms: ARM A: intensive nutritional intervention

SUMMARY:
The present trial aims to compare the effectiveness of an "intensive" vs a "standard" nutritional intervention on body weight regulation and some metabolic parameters in women on adjuvant/neoadjuvant therapy for breast cancer.

DETAILED DESCRIPTION:
The effectiveness of an "intensive" versus "non-intensive" dietary intervention will be assessed in 120 patients on adjuvant therapy for breast cancer (BC) in a prospective, randomized controlled study for a total of 3 years. The eligibility of participants will be verified according to the inclusion/exclusion criteria at the screening visit; therefore, after a detailed explanation of the study protocol, Informed Consent will be signed. After the recruitment, subjects will be randomized into an "intensive" (ARM A) and "non-intensive" (ARM B) dietary intervention group. After the 6 month treatment period, patients will be followed up for the following 18 months.

ARM A: Visits will be set up monthly in order to assess body weight, waist circumference, diet compliance (etc...) for all period of the BC adjuvant treatment (6 months).

ARM B: Visits will be set up only at the baseline, after 6 months namely at the end.

No drug treatment will be given to patients during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old
* BMI < 30 kg/m2
* Caucasians
* Histological diagnosis of invasive breast cancer
* Starting an adjuvant systemic treatment for breast cancer
* Available past medical history
* Informed consent to participate to the study

Exclusion Criteria:

* Metastatic disease
* BMI >30 kg/m2
* Presence of a serious medical condition that could alter food absorption or prognosis
* Refusal to provide informed consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Body weight control | 12 months
  To investigate the effects of an intensive nutritional intervention on Body weight control (defined as weight changes ≤+5% of the initial body weight) at 12 months after the beginning of systemic treatment.

SECONDARY OUTCOMES:
Body weight | From enrollment to 6, 12 and 24 months
  To evaluate the effects of an intensive nutritional intervention at 6, 12 and 24 months after the beginning of systemic treatment on:
  - Body weight (Kg)
Body Mass Index (BMI) | From enrollment to 6, 12 and 24 months
  Body Mass Index (BMI)
  Kg/m2
Body composition | From enrollment to 6, 12 and 24 months
  Body composition
  Body composition will be assessed with Bio-impedance analysis (BIA) at 50 kilohertz (kHz) (Human Im Plus II, Medica) at room temperature of 22-25 °C.
Resting energy expenditure (REE) | From enrollment to 6, 12 and 24 months
  Resting energy expenditure (REE)
  Resting Energy Expenditure will be measured (MREE) by indirect calorimetry using a canopy system (V max29, Sensor Medics, U.S.A.) at an ambient temperature of 23-25 °C.
Quality of life (QoL) | From enrollment to 6,12 and 24 months
  Quality of life (QoL)
  Assessed with European Organisation For Research And Treatment Of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 (version 3.0)
  The EORTC QLQ-C30 questionnaire yields scores ranging from 0 to 100 for each domain. For functional scales and the global health status/QoL scale, higher scores indicate better functioning or quality of life, meaning a higher score represents a better outcome. In contrast, for symptom scales and single items (e.g., fatigue, pain, nausea), higher scores indicate more severe symptoms, meaning a higher score reflects a worse outcome.
Change from Baseline in the Mean concentration of Fasting glucose | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -Fasting glucose (mg/dl)
Change from Baseline in the Mean concentration of Serum insulin (mg/dl) | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -serum insulin concentration (mg/dl)
Change from Baseline in the Mean concentration of C-peptide (ng/ml) | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  * C-peptide (ng/ml)
Change from Baseline in the Mean concentration of glycosylated haemoglobin | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  * glycosylated haemoglobin (%)
Change from Baseline in the Mean concentration of total cholesterol | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  * total cholesterol (mg/dl)
Change from Baseline in the Mean concentration of HDL cholesterol | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -HDL cholesterol (mg/dl)
Change from Baseline in the Mean concentration of LDL cholesterol | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -LDL cholesterol (mg/dl)
Change from Baseline in the Mean concentration of triglycerides | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -triglycerides (mg/dl)
Change from Baseline in the Mean concentration of urea | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -urea (mg/dl)
Change from Baseline in the Mean concentration of creatinine | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -creatinine (mg/dl)
Change from Baseline in the Mean concentration of urate | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -urate (mg/dl)
Change from Baseline in the Mean concentration of Aspartate Amino Transaminase | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  - Aspartate Amino Transaminase (AST) (U/L)
Change from Baseline in the Mean concentration of Alanine AminoTransferase | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  - Alanine AminoTransferase (ALT) (U/L)
Change from Baseline in the Mean concentration of Gamma-Glutamyl Transferase | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -Gamma-Glutamyl Transferase (GGT) (U/L)
Change from Baseline in the Mean concentration of Alkaline Phosphatase | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  - Alkaline Phosphatase (ALP) (U/L)
Change from Baseline in the Mean concentration of erythrocytes Sedimentation Rate | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  - Erythrocyte Sedimentation Rate (ESR) (U/L)
Change from Baseline in the Mean concentration of C-reactive protein | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -C-reactive protein (PCR) (U/L)
Change from Baseline in the Mean concentration of Thyroid-stimulating hormone | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -Thyroid-stimulating hormone (TSH) (mUI/L)
Change from Baseline in the Mean concentration of Free Triiodothyronine | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -Free Triiodothyronine (FT3) (pg/ml)
Change from Baseline in the Mean concentration of Free thyroxine | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -Free thyroxine (FT4) (pg/ml)
Change from Baseline in the Mean concentration of vitamin D | From enrollment to 6,12 and 24 months
  Serum metabolic variables (concentration)
  -vitamin D (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
Past medical history, clinico-pathological informations, anthropometric variables, survival status.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT07044791/Prot_SAP_000.pdf
  • Informed Consent Form: English version (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT07044791/ICF_001.pdf